CLINICAL TRIAL: NCT05009537
Title: Optical Genome Mapping in Hematological Malignancies
Acronym: CARTOGEN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CARTOGEN - 29BRC21.0211
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: MDS; ALL; Other Hematologic Malignant Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — fresh cells from bone marrow frozen cells frmp bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establish the diagnostic potential of optical genome mapping in patients with suspected hematologic cancer

ELIGIBILITY:
Inclusion Criteria:

* Minor/Major Patients
* Patients with suspected hemopathies for whom we receive a sample for diagnosis in the chromosomal genetics laboratory or for whom a diagnosis of hemopathy has already been made.
* No objection made or consent given

Exclusion Criteria:

* Patients under judicial protection (guardianship, curatorship, ...),
* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected hemopathies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Establish the diagnostic potential of optical genome mapping in patients with suspected hematologic cancer | 2021-2026
  identification of anomalies by mapping identical to those identified by combining conventional cytogenetics and FISH.

SECONDARY OUTCOMES:
identification of new chromosomal abnormalities of clinical relevance. | 2021-2026
identification of new chromosomal anomalies involved in oncogenic pathways | 2021-2026

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHRU de Brest, Brest
  - CH Morlaix, service d'hémato clinique, Morlaix
  - CHIC, service d'hémato clinique, Quimper
  - CH St Brieuc, service d'hémato clinique, Saint-Brieuc

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. requestors will be required to sign and complete a data access agreement